CLINICAL TRIAL: NCT04598906
Title: Comparison of the Effectiveness of the Virtual Environment in Cognitive Rehabilitation With Standard Rehabilitation Methods in Patients With Schizophrenia and in Patients With Major Depressive Disorder
Brief Title: Ecologically Valid Virtual Tasks vs Paper-pencil Methods in Cognitive Rehabilitation in Patients With Schizophrenia and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Responsible Party: Principal Investigator, Adéla Plechatá, researcher, PhD student, National Institute of Mental Health, Czech Republic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VRremediation
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia; Depression; Cognitive Impairment
Keywords: cognitive deficit; schizophrenia; major depressive disorder; virtual environment; cognitive rehabilitation
MeSH Terms: conditions — Schizophrenia; Depression; Cognitive Dysfunction; Cognition Disorders; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual environment rehabilitation - Paper-pencil rehabilitation (Experimental): The participants in this arm completes Virtual environment rehabilitation as the first condition and then crossover to Paper-pencil rehabilitation.
  Interventions: Behavioral: Virtual environment rehabilitation; Behavioral: Paper-pencil rehabilitation
- Paper-pencil rehabilitation - Virtual environment rehabilitation (Experimental): The participants in this arm completes Paper-pencil rehabilitation as the first condition and then crossover to Virtual environment rehabilitation.
  Interventions: Behavioral: Virtual environment rehabilitation; Behavioral: Paper-pencil rehabilitation

INTERVENTIONS:
Behavioral: Virtual environment rehabilitation — The participants attended 10-15 computer sessions during 6-12 weeks. Each session lasted 30 minutes and consisted of the set of virtual environment tasks (Shooting Range,Virtual Supermarket Shopping Task and Objects). Shooting range demands differentiation of targets from non-targets and focuses on training of selective attention, psychomotor speed and inhibition control. Virtual Supermarket Shopping requires memorizing the shopping list and searching for products in the supermarket area. Objects requires memorizing of the spatial and temporal context while searching for objects.
Behavioral: Paper-pencil rehabilitation — The participants in the paper-pencil rehabilitation attended 10-15 paper pencil sessions for 6-12 weeks. Each session lasted 45 minutes. Each paper-pencil session starts with a warm-up game. The session continues with a set of paper-pencil tasks focused on attention, fine motor skills, recall, short-term and long-term memory, verbal fluency, visual search, cognitive flexibility, abstraction and executive functions, numerical abilities. The tasks are adapted according to the participant´s abilities.

SUMMARY:
Schizophrenia is heterogeneous and often disabling a disease that affects 1% of the population. Current psychopharmacological treatment significantly eliminates the presence of positive symptoms (especially delusions and hallucinations) and partly also negative symptoms (social withdrawal or abulia). In contrast, the cognitive deficits associated both with schizophrenia and depression are only limitedly influenced by pharmacological treatment.The cognitive impairment represents an important part of schizophrenia symptomatology and it has a severe negative impact on patients' quality of life. In depression is the impairment milder but still significantly contributes to patients' daily functioning. The profound deficit was repeatedly documented in the area of declarative and working memory. In this study, we study the effectiveness of virtual environment rehabilitation program focused on declarative memory, working memory and attention in comparison to standard paper-pencil rehabilitation led by an occupational therapist.

DETAILED DESCRIPTION:
This study compares effectiveness of the virtual environment cognitive rehabilitation program with standard paper-pencil approach in within-subject design.

Participants with a diagnosis of schizophrenia, schizoaffective disorder or major depressive disorder will undergo a baseline assessment of cognition.

The participants will be at the baseline randomly assigned to each condition: virtual environment rehabilitation or paper-pencil rehabilitation. Then they will participate in 10-15 sessions (30-45 minutes) once or twice a week.

All participants will undergo retest assessment of cognition.

After completion of the first program the participants will be assigned to the different condition: to paper-pencil or virtual environment rehabilitation. After 10-15 sessions in the second condition the participants will once more undergo retest assessment of cognition.

Within-subject design is an effective tool in the development of scientifically proven treatment tools. This approach allows to obtain reliable information about the effectiveness of the method and to examine the influences of other variables (Steingrimsdottir and Arntzen 2015). This study will allow to get credible information on the importance of using the virtual environment in the context of cognitive rehabilitation in patients with schizophrenia and depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia and other primary psychotic disorders or diagnosis of major depressive disorder according to International Classification of Diseases-11

Exclusion Criteria:

* Severe visual impairment
* Age over 60 years
* Diagnosis of other psychiatric disorder than schizophrenia or major depressive disorder
* Physical handicap preventing the participant from participating in virtual environment training
* Refusal to sign an informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Cognitive abilities measured by The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline, 6-12 weeks, 12-24 weeks

SECONDARY OUTCOMES:
Item performance in Virtual Supermarket Shopping Task | Baseline, 6-12 weeks
  The data from individual sessions with Virtual Supermarket Shopping Task will be analyzed to see participants' progress. The variable item performance will be used = number of items to remember/ correctly collected items.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Center, Fryštát, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steingrimsdottir HS, Arntzen E. On the utility of within-participant research design when working with patients with neurocognitive disorders. Clin Interv Aging. 2015 Jul 23;10:1189-99. doi: 10.2147/CIA.S81868. eCollection 2015. PMID 26229453